CLINICAL TRIAL: NCT00001068
Title: Influence of Risk Status for Disease Progression on the Response to Antiretroviral Interventions: A Follow-up Study to ACTG 175
Brief Title: A Study of Disease Progression and Anti-HIV Treatments
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: ACTG 303; 11278 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Zalcitabine; Didanosine; Drug Therapy, Combination; AIDS-Related Complex; Antiviral Agents; Zidovudine; Lamivudine
MeSH Terms: conditions — HIV Infections; AIDS-Related Complex | interventions — Lamivudine

INTERVENTIONS:
Drug: Lamivudine

SUMMARY:
To determine the influence of virus load, CD4 count, biologic phenotype, and presence of symptomatic disease on the response of HIV-infected patients to a new therapeutic regimen. PER AMENDMENT 8/27/96: To extend the availability of currently assigned ACTG 303 treatment for 6 months.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Prior participation on protocol ACTG 175.

PER AMENDMENT 8/27/96:

* Patients must be on study/on treatment at the time the protocol study treatment is extended.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 210
Dates: Study Completion 1998-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (41):
- United States (39):
  - Alabama Therapeutics CRS, Birmingham, Alabama
  - USC CRS, Los Angeles, California
  - UCLA CARE Center CRS, Los Angeles, California
  - Stanford CRS, Palo Alto, California
  - Ucsd, Avrc Crs, San Diego, California
  - Ucsf Aids Crs, San Francisco, California
  - Santa Clara Valley Med. Ctr., San Jose, California
  - San Mateo County AIDS Program, Stanford, California
  - Harbor-UCLA Med. Ctr. CRS, Torrance, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Univ. of Miami AIDS CRS, Miami, Florida
  - Emory Univ. Hemophilia Program Office, Atlanta, Georgia
  - Northwestern University CRS, Chicago, Illinois
  - Cook County Hosp. CORE Ctr., Chicago, Illinois
  - Rush Univ. Med. Ctr. ACTG CRS, Chicago, Illinois
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - Tulane Hemophilia Treatment Ctr., New Orleans, Louisiana
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland
  - Massachusetts General Hospital ACTG CRS, Boston, Massachusetts
  - Bmc Actg Crs, Boston, Massachusetts
  - Beth Israel Deaconess - East Campus A0102 CRS, Boston, Massachusetts
  - Beth Israel Deaconess Med. Ctr., ACTG CRS, Boston, Massachusetts
  - University of Minnesota, ACTU, Minneapolis, Minnesota
  - St. Louis ConnectCare, Infectious Diseases Clinic, St Louis, Missouri
  - Washington U CRS, St Louis, Missouri
  - Univ. of Nebraska Med. Ctr., Durham Outpatient Ctr., Omaha, Nebraska
  - SUNY - Buffalo, Erie County Medical Ctr., Buffalo, New York
  - Beth Israel Med. Ctr. (Mt. Sinai), New York, New York
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Cornell University A2201, New York, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - Unc Aids Crs, Chapel Hill, North Carolina
  - Carolinas HealthCare System, Carolinas Med. Ctr., Charlotte, North Carolina
  - Regional Center for Infectious Disease, Wendover Medical Center CRS, Greensboro, North Carolina
  - Univ. of Cincinnati CRS, Cincinnati, Ohio
  - Case CRS, Cleveland, Ohio
  - The Ohio State Univ. AIDS CRS, Columbus, Ohio
  - Hosp. of the Univ. of Pennsylvania CRS, Philadelphia, Pennsylvania
  - University of Washington AIDS CRS, Seattle, Washington
- Puerto Rico-AIDS CRS, San Juan, Puerto Rico
- Mbeya Med. Research Program, Mbeya Referral Hosp. CRS, Mbeya, Tanzania

REFERENCES:
- [Background] Albrecht MA, Hughes MD, Liou SH, Katzenstein DA, Murphy R, Balfour HH, Para MF, Valdez H, Hammer SM; ACTG 303 Study Team. Effect of lamivudine in HIV-infected persons with prior exposure to zidovudine/didanosine or zidovudine/zalcitabine. AIDS Res Hum Retroviruses. 2000 Sep 20;16(14):1337-44. doi: 10.1089/08892220050140883. PMID 11018853